CLINICAL TRIAL: NCT06726954
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation Therapy in Neuropathic Pain Associated With Spinal Cord Injury; Randomized Controlled Trial
Brief Title: Repetitive Transcranial Magnetic Stimulation Therapy in Spinal Cord Injury Related Neuropathic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Nuran Eyvaz, Assistant Professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMSSCINP
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
Keywords: Transcranial Magnetic Stimulation; Spinal Cord Injury; Neuropathic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First Group (Experimental): High-frequency real-time rTMS protocol It was planned to apply the dorsolateral prefrontal cortex daily at a frequency of 10 Hz for 20 sessions.
  Interventions: Device: High-frequency real-time rTMS DLPF cortex protocol
- Second Group (Experimental): High-frequency real-time rTMS protocol It was planned to apply the M1 motor cortex daily at a frequency of 10 Hz for 20 sessions.
  Interventions: Device: High-frequency real-time rTMS M1 motor cortex protocol
- Third Group (Sham Comparator): Sham rTMS Protocol It was planned to apply daily sham rTMS for 20 sessions.
  Interventions: Device: Sham rTMS Protocol

INTERVENTIONS:
Device: High-frequency real-time rTMS DLPF cortex protocol — It was planned to apply the dorsolateral prefrontal cortex daily for 20 sessions.Along with the daily rTMS session, participants will continue to use the medications in the medical treatment at the same effective dose and no dose changes will be made during the treatment.
  Arms: First Group
Device: High-frequency real-time rTMS M1 motor cortex protocol — It was planned to apply the M1 motor cortex daily for 20 sessions.Along with the daily rTMS session, participants will continue to use the medications in the medical treatment at the same effective dose and no dose changes will be made during the treatment.
  Arms: Second Group
Device: Sham rTMS Protocol — It was planned to apply the daily for 20 sessions.Along with the daily rTMS session, participants will continue to use the medications in the medical treatment at the same effective dose and no dose changes will be made during the treatment.
  Arms: Third Group

SUMMARY:
The aim of our study is to investigate the effect of different protocols of high-frequency Repetitive Transcranial Magnetic Stimulation (rTMS) therapy added to the rehabilitation program on neuropathic pain,depression, quality of life and quality of sleep compared to each other and placebo group in participants with spinal cord injury.

DETAILED DESCRIPTION:
Spinal cord injury is a disability that causes the loss of many functions for example motor,sensory and autonomic functions in the body. Neuropathic pain is a common problem in participants with spinal cord injury. Many treatment options have been offered for a debilitating condition that has major negative effects on participant's quality of life but provides limited effects and many secondary effects. There is evidence for neuromodulation techniques to improve many pain conditions, such as neuropathic pain. One innovative method for neuropathic pain management, rTMS, is a non-invasive neuromodulation intervention with a low risk of side effects that works by altering brain activity. While most studies to date have mainly targeted the primary motor cortex (M1), fewer studies have reported analgesic effects after stimulation of other cortical areas such as the dorsolateral prefrontal cortex (DLPFC).

The initial assessment will include answering questionnaires: Brief Pain Inventory, Neuropathic Pain Symptom Inventory(NPSI), International Spinal Cord Injury Pain Basic Data Set (ISCIPBDS) self-report version, Patient Catastrophizing Scale(PCS), Beck Depression Inventory,Quality of Life Index Spinal Cord Injury v3 (QLI-SCI), Pain Catastrophizing Scale (PCS),Pittsburgh Sleep Quality Index and previous medication and treatment questionnaires.Participants will be asked to complete the above-mentioned questionnaires post-rTMS treatment and at 2 months after their last rTMS treatment.

TMS Protocol: Participants will undergo high frequency rTMS sessions 5 days a week for 4 weeks (20 treatments total). Daily rTMS sessions will include at a frequency of 10 Hz, treatment intensity will be applied at 120% of the participants resting motor threshold (RMT). A RMT is the minimal intensity required to evoke a motor evoked potential and will be obtained by administering single-pulse TMS to the left motor cortex participant a will be seated in a comfortable chair or their wheelchair for each rTMS session.

Participants with spinal cord injury receiving rTMS in DLPFC or M1 protocol in addition to neurological rehabilitation will be compared with the sham rTMS group in terms of neuropathic pain, sleep quality, depression and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Aged 18-75 years Physician-diagnosed spinal cord injury for at least 3-months Neuropathic pain for at least 3-months Pain not attributable to any other conditions

Exclusion Criteria:

* Having an important comorbid disease such as severe heart disease (aortic stenosis, angina, hypertrophic cardiomyopathy, uncontrolled hypertension,arrhythmia, pacemaker)
* Neurodegenerative disease
* Epilepsy
* History of antiepileptic drug use
* Cognitive dysfunction
* Lower extremity peripheral nerve injury
* Increased intracranial pressure or uncontrolled migraine
* Infection on the skin in the application area.
* Having a brain lesion or a history of drug use that will affect the seizure threshold.

Any TMS-related contraindications, for example:

* Pacemaker
* Metallic implant
* Previous seizure
* Psychiatric disorders (excluding depression and anxiety)
* Malignancy
* Current pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Brief Pain Inventory-Short Form (BPI-SF) at 1. and 2 months. | To be assessed at baseline, after rTMS treatment (1-month) and 2-months after rTMS treatment.
  The Brief Pain Inventory Short Form (SPI-SF) is designed to examine pain in terms of sensory (pain intensity) and impact on daily functioning. The BPI-SF consists of two parts. The first part assesses the severity of worst, mildest, average and momentary pain using a numerical rating scale (NRS; 0-10). A response of 0 indicates "no pain at all" and a response of 10 indicates "the most severe pain imaginable". The second part consists of seven questions assessing how much pain affects daily functioning, including general activity and enjoyment of life. A response of 0 indicates "not at all affected" and a response of 10 indicates "completely affected". The total score ranges from 0-70. Higher scores indicate worsening symptoms.

SECONDARY OUTCOMES:
Change from baseline International Spinal Cord Injury Pain Basic Data Set (ISCIPBDS) self-report version at 1. and 2 months. | To be assessed at baseline, after rTMS treatment (1-month) and 2-months after rTMS treatment.
  Pain profile, including location, intensity, and interference over the past 7 days will be assessed using the ISCIPBDS self-report tool. All variables are rated on a scale ranging from 0 (no pain at all) to 10(the most severe pain imaginable).Higher scores indicate higher pain intensity.
Change from baseline Quality of Life Index Spinal Cord Injury version (QLI-SCI) at 1. and 2 months. | To be assessed at baseline, after rTMS treatment (1-month) and 2-months after rTMS treatment.
  Quality of life and satisfaction with aspects of quality of life will be assessed using the QLI-SCI instrument. This questionnaire focuses on the categories of health and functioning, social and economic, psychological/spiritual, and family. All variables are rated on a scale ranging from 0 (completely dissatisfied) to 10(completely satisfied) with a total of 40 points. Higher scores indicates better quality of life.
Change from baseline Pain Catastrophizing Scale (PCS) at 1. and 2 months. | To be assessed at baseline, after rTMS treatment (1-month) and 2-months after rTMS treatment.
  Pain experience will be assessed using the PCS. Participants are asked to rate how much they agree with the listed thoughts and feelings they may have when experiencing pain from 0 (not at all) to 4 (all the time). The total score ranges from 0-52. Higher scores indicate increase level of catastrophizing.
Change from baseline Beck Depression Inventory (BDI) Scores at 1. and 2 months. | To be assessed at baseline, after rTMS treatment (1-month) and 2-months after rTMS treatment.
  Validated measure of clinical depression symptoms to quantify and track mood over time. Scores index depression severity and range from 0-63: 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.Total score is 63. Higher scores indicates depressive mood.
Change in the Patient's Global Impression of Change (PGIC) observed at 1 month and 2 months. | To be assessed after rTMS treatment (1-month) and 2-months after rTMS treatment.
  Standardized assessment to assess participants overall impression of improvement. Scores range from 1 to 7, with 1 representing "no change" and 7 representing "a great deal better"
Change from baseline Neuropathic Pain Symptom Inventory (NPSI) at 1.and 2 months. | To be assessed at baseline, after rTMS treatment (1-month) and 2-months after rTMS treatment.
  An 11-point NRS assess average neuropathic pain severity over the last week. The scale ranged from 0 to 10, with 0 representing "no pain" and 10 representing "the most intense pain imaginable". The NPSI is comprised of five subscales: burning spontaneous pain (burning), pressing spontaneous pain (pressing), paroxysmal pain (paroxysmal), evoked pain (evoked), and paresthesia/dysesthesia. Full scale from 0-10, with higher score indicating more symptom.
Change from baseline Pittsburgh Sleep Quality Index (PSQI) at 1. and 2 months. | To be assessed at baseline, after rTMS treatment (1-month) and 2-months after rTMS treatment.
  The Pittsburgh Sleep Quality Index (PSQI) is an 18-item questionnaire that assesses sleep quality and disturbances over the past month. The investigators will use the 3-factor scoring, which has been shown to have superior psychometric properties.
  The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Change from baseline Modified Ashworth Scale (MAS) at 1. and 2 months. | To be assessed at baseline, after rTMS treatment (1-month) and 2-months after rTMS treatment.
  Modified Ashworth Scale (MAS) will measure spasticity in the limbs. Higher scores represent spasticity or increased resistance to passive movement. All variables are rated on a scale ranging from 0 to 5: 0 means no increase in muscle tone (better outcome) and 5 means rigid (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Nuran Eyvaz, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Background] Attal N, Poindessous-Jazat F, De Chauvigny E, Quesada C, Mhalla A, Ayache SS, Fermanian C, Nizard J, Peyron R, Lefaucheur JP, Bouhassira D. Repetitive transcranial magnetic stimulation for neuropathic pain: a randomized multicentre sham-controlled trial. Brain. 2021 Dec 16;144(11):3328-3339. doi: 10.1093/brain/awab208. PMID 34196698
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Saleh C, Ilia TS, Jaszczuk P, Hund-Georgiadis M, Walter A. Is transcranial magnetic stimulation as treatment for neuropathic pain in patients with spinal cord injury efficient? A systematic review. Neurol Sci. 2022 May;43(5):3007-3018. doi: 10.1007/s10072-022-05978-0. Epub 2022 Mar 3. PMID 35239053